CLINICAL TRIAL: NCT02036918
Title: Evaluation of Lymph Node Metastases in Men Undergoing Treatment With Sipuleucel-T for Metastatic Castrate-resistant Prostate Cancer
Brief Title: Dendreon Lymph Node Biopsy in Metastatic Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00047231
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: castrate resistant prostate cancer; metastatic; sipuleucel-T; lymphadenectomy; Excisional lymph node biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — sipuleucel-T; Sentinel Lymph Node Biopsy; Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Pre-treatment control group will be randomized to immediate lymph node biopsy followed by sipuleucel-T immunotherapy.
  Interventions: Drug: Sipuleucel-T; Procedure: Lymph Node Biopsy
- Arm B (Experimental): Post-treatment experimental group will be randomized to immediate sipuleucel-T immunotherapy followed by lymph node biopsy.
  Interventions: Drug: Sipuleucel-T; Procedure: Lymph Node Biopsy

INTERVENTIONS:
Drug: Sipuleucel-T
  Other Names: Provenge
Procedure: Lymph Node Biopsy
  Other Names: lymphadenectomy; lymph node dissection; excisional lymph node biopsy

SUMMARY:
This study aims to evaluate patients with metastatic castrate-resistant prostate cancer (mCRPC) undergoing treatment with sipuleucel-T for evidence of treatment-associated immune activation in lymph nodes and peripheral blood.

DETAILED DESCRIPTION:
This is a pilot study of mCRPC patients planning to undergo therapy with sipuleucel-T immunotherapy. Consenting patients will be randomized 3:1 between immediate sipuleucel-T immunotherapy followed by lymph node biopsy (the post-treatment experimental group) or immediate lymph node biopsy followed by sipuleucel-T immunotherapy (the pre-treatment control group). Peripheral blood will be collected before, during, and after treatment with sipuleucel-T and evaluated for evidence of sipuleucel-T induced immune activation. Lymph nodes collected at biopsy will also be evaluated for evidence of sipuleucel-T induced immune activation. Patients will be followed for 3 months for safety and 6 months for disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. ECOG performance status 0 or 1
3. Life expectancy of ≥ 6 months
4. Minimally-symptomatic or asymptomatic, castrate-resistant metastatic prostate cancer, as evidenced by all of the following:

   1. Histologically-confirmed diagnosis of adenocarcinoma of the prostate
   2. Evidence of adequate androgen deprivation, as evidence by one of the following:

      * Bilateral orchiectomy
      * Ongoing LHRH agonist (e.g. leuprolide, goserelin) and serum testosterone <50 ng/dl
      * Ongoing LHRH antagonist (e.g. degarelix) and serum testosterone <50 ng/dl
   3. Evidence of prostate cancer resistance to castration, as evidenced by one of the following:

      * 2 consecutive PSA levels that are ≥ 50% above the PSA nadir achieved on ADT and obtained at least 1 week apart
      * CT or MRI based evidence of disease progression (soft tissue or nodal) according to PCWG2 criteria or RECIST 1.1 criteria, or at least 1 new bone scan lesion as compared to the most immediate prior radiologic studies.
   4. Presence of non-visceral metastases on imaging
   5. Absence of major symptoms directly attributable to prostate cancer, with the following permissible exceptions:

      * Ureteral obstruction secondary to pelvic or retroperitoneal lymphadenopathy
      * Bladder outlet obstruction secondary to locally recurrent prostate cancer
5. Radiographic evidence of lymphadenopathy, defined as a lymph node greater than 1 cm in diameter on axial imaging (CT or MRI or PET/CT)
6. Adequate laboratory parameters
7. A minimum of 4 weeks from any major surgery prior to registration. Coincident standard of care surgery with the research biopsy is permitted during the study.

Exclusion Criteria:

1. Prior treatment with sipuleucel-T
2. Allergy to any component of sipuleucel-T
3. Inability to undergo leukapheresis
4. History of neuroendocrine variants of prostate cancer, including small cell carcinoma of the prostate
5. Extensive prior surgery/radiation present that would render the biopsy highly complex and the risk of intraoperative injury high
6. Any chronic medical condition requiring daily corticosteroids or other immunosuppressants
7. Solid organ transplantation requiring immunosuppression
8. Visceral (e.g. lung, liver) metastases
9. Known brain metastases
10. History of spinal cord compression
11. Untreated/unstabilized pathologic long bone fractures
12. Other malignancy, except non-melanoma skin cancer, with a ≥ 30% probability of recurrence within 24 months
13. Administration of any investigational therapeutic within 30 days of registration
14. Any condition which, in the opinion of the investigator, would preclude participation in this trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
anti-PA2024 immune response in lymph node-derived leukocytes | Lymph node biopsy, approximately 10 weeks
  Proportion of patients with lymph node-derived leukocytes showing anti-PA2024 activity as measured by IFNγ ELISPOT
anti-PAP immune response in lymph node-derived leukocytes | Lymph node biopsy, approximately 10 weeks
  Proportion of patients with lymph node-derived leukocytes showing anti-PAP activity as measured by IFNγ ELISPOT
anti-PA2024 immune response in PBMCs | Baseline
  Proportion of patients with PBMC samples showing anti-PA2024 activity as measured by IFNγ ELISPOT at each time point
anti-PAP immune response in PBMCs | Baseline
  Proportion of patients with PBMC samples showing anti-PAP activity as measured by IFNγ ELISPOT at each time point
anti-PA2024 immune response in PBMCs | Prior to sipuleucel-T infusion 2, approximately 6 weeks
  Proportion of patients with PBMC samples showing anti-PA2024 activity as measured by IFNγ ELISPOT at each time point
anti-PAP immune response in PBMCs | Prior to sipuleucel-T infusion 2, approximately 6 weeks
  Proportion of patients with PBMC samples showing anti-PAP activity as measured by IFNγ ELISPOT at each time point
anti-PA2024 immune response in PBMCs | Prior to sipuleucel-T infusion 3, approximately 8 weeks
  Proportion of patients with PBMC samples showing anti-PA2024 activity as measured by IFNγ ELISPOT at each time point
anti-PAP immune response in PBMCs | Prior to sipuleucel-T infusion 3, approximately 8 weeks
  Proportion of patients with PBMC samples showing anti-PAP activity as measured by IFNγ ELISPOT at each time point
anti-PA2024 immune response in PBMCs | 2 weeks after the last sipuleucel-T infusion
  Proportion of patients with PBMC samples showing anti-PA2024 activity as measured by IFNγ ELISPOT at each time point
anti-PAP immune response in PBMCs | 2 weeks after the last sipuleucel-T infusion
  Proportion of patients with PBMC samples showing anti-PAP activity as measured by IFNγ ELISPOT at each time point
anti-PA2024 immune response in PBMCs | 3 months post-treatment
  Proportion of patients with PBMC samples showing anti-PA2024 activity as measured by IFNγ ELISPOT at each time point
anti-PAP immune response in PBMCs | 3 months post-treatment
  Proportion of patients with PBMC samples showing anti-PAP activity as measured by IFNγ ELISPOT at each time point
anti-PA2024 immune response in PBMCs | 6 months post-treatment
  Proportion of patients with PBMC samples showing anti-PA2024 activity as measured by IFNγ ELISPOT at each time point
anti-PAP immune response in PBMCs | 6 months post-treatment
  Proportion of patients with PBMC samples showing anti-PAP activity as measured by IFNγ ELISPOT at each time point

SECONDARY OUTCOMES:
Serum anti-PA2024 antibody level | Baseline, up to 6 months post-treatment
  Describe any relationship between the magnitude of sipuleucel-T induced leukocyte activation observed in tumor-bearing lymph nodes with systemic (i.e. peripheral blood) studies of sipuleucel-T-induced immune activation
serum anti-PAP antibody level | Baseline, up to 6 months post-treatment
  Describe any relationship between the magnitude of sipuleucel-T induced leukocyte activation observed in tumor-bearing lymph nodes with systemic (i.e. peripheral blood) studies of sipuleucel-T-induced immune activation

CONTACTS AND LOCATIONS:
Overall Officials: Brant Inman, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States